CLINICAL TRIAL: NCT04922489
Title: Clinical Outcome of Dentsply Sirona EV Implants: A Retrospective Study of 500 Implants With 6-year Follow-up
Brief Title: Clinical Outcome of Dentsply Sirona EV Implants
Status: Completed | Type: Observational
Sponsor: Aula Dental Avanzada (Other)
Responsible Party: Principal Investigator, Guillem Esteve-Pardo, Principal Investigator, Aula Dental Avanzada
Other Study IDs: RETRODSI
Record Dates: First submitted 2021-06-03; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Dental Implants
Keywords: Dental Implant; Complication; Astra Tech EV
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Astra Tech EV: Patients who has receive Astra Tech dental implant system placement.
  Interventions: Procedure: Dental implant placement

INTERVENTIONS:
Procedure: Dental implant placement — Dental implant placemente on edentulous jaw.
  Other Names: Implant surgery; Implant prosthesis

SUMMARY:
Retrospective observational study of 500 implants placed between 2014 and 2020 of the same dental implant system (AstraTech Implant System EV, Dentsply Implants, Mölndal, Sweden).

DETAILED DESCRIPTION:
The purpose of this study is to assess the cumulative survival, success and complications rates obtained with the use of AstraTech Implant System EV in one clinical center from market launch to 2020

All clinical records of patients with this implant system will be collected and the following data will be recorded:

Patient gender Date of placement Dimensions and location of implant(s) placed Type of implantation Design of the implant-supported dental prosthesis, single or partial, screw-retained or cemented Date of last radiographic control Type of biological and/or mechanical complications that occurred In biological complications, presence or absence of inflammatory signs and presence or absence of peri-implant bone loss.

For mechanical complications, screw loosening, porcelain fracture, fracture of the prosthetic abutment or fracture of the implant.

Date of explantation if present

The mean, standard deviation (SD), and percentage will be calculated for all recorded parameters.

A life table will be made with cumulative survival and success rate (CSR), according to Kaplan-Meier analysis. Correlations and regression analysis will be performed to assess the influence of the variables on the outcomes

Conclusions will be drawn based on the results obtained.

ELIGIBILITY:
Inclusion Criteria:

All patients who receive Astra Tech EV dental implant system placement.

Exclusion Criteria:

None

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Male or female
Study Population: All patients who receive Astra Tech EV dental implant system placement al private practice in Clinica Dental Esteve in Alicante (Spain).
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Implant Success | through study completion, a maximum of 5 year
  Dental Implants in function with no complications events
Implant survival | through study completion, a maximum of 5 year
  Dental Implants in function with any complications events

SECONDARY OUTCOMES:
Biological complications | through study completion, a maximum of 5 year
  Dental implant treatment with some biological complication
Mechanical complications | through study completion, a maximum of 5 year
  Dental implant treatment with some mechanical complication

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Esteve-Pardo, DDS, Principal Investigator — Aula Dental Avanzada
Locations (1):
- Clínica Dental Esteve, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norton MR, Astrom M. The Influence of Implant Surface on Maintenance of Marginal Bone Levels for Three Premium Implant Brands: A Systematic Review and Meta-analysis. Int J Oral Maxillofac Implants. 2020 Nov/Dec;35(6):1099-1111. doi: 10.11607/jomi.8393. PMID 33270049
- [Background] Astrand P, Engquist B, Dahlgren S, Grondahl K, Engquist E, Feldmann H. Astra Tech and Branemark system implants: a 5-year prospective study of marginal bone reactions. Clin Oral Implants Res. 2004 Aug;15(4):413-20. doi: 10.1111/j.1600-0501.2004.01028.x. PMID 15248875
- [Background] Derks J, Schaller D, Hakansson J, Wennstrom JL, Tomasi C, Berglundh T. Effectiveness of Implant Therapy Analyzed in a Swedish Population: Prevalence of Peri-implantitis. J Dent Res. 2016 Jan;95(1):43-9. doi: 10.1177/0022034515608832. PMID 26701919
- [Background] Chae SW, Kim YS, Lee YM, Kim WK, Lee YK, Kim SH. Complication incidence of two implant systems up to six years: a comparison between internal and external connection implants. J Periodontal Implant Sci. 2015 Feb;45(1):23-9. doi: 10.5051/jpis.2015.45.1.23. Epub 2015 Feb 25. PMID 25722923
- [Background] Choi NH, Yoon HI, Kim TH, Park EJ. Improvement in Fatigue Behavior of Dental Implant Fixtures by Changing Internal Connection Design: An In Vitro Pilot Study. Materials (Basel). 2019 Oct 7;12(19):3264. doi: 10.3390/ma12193264. PMID 31591290
- [Background] Toia M, Galli S, Cecchinato D, Wennerberg A, Jimbo R. Clinical Evidence of OsseoSpeed EV Implants: A Retrospective Study and Characterization of the Newly Introduced System. Int J Periodontics Restorative Dent. 2019 November/December;39(6):863-874. doi: 10.11607/prd.2549. Epub 2017 Aug 23. PMID 28834532